CLINICAL TRIAL: NCT02291432
Title: Muscle Cell Mediated Therapy for Stress Urinary Incontinence in Males Following Prostate Surgery: An Investigation of Cook MyoSite Autologous Muscle Derived Cells
Brief Title: Autologous Cell Therapy for Stress Urinary Incontinence in Males Following Prostate Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cook MyoSite (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-11
Record Dates: First submitted 2014-11-11; First posted 2014-11-14 (Estimated); Results first posted 2021-10-26 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Urinary Incontinence; Stress; Urination Disorders; Urologic Diseases; Lower Urinary Tract Symptoms; Urological Manifestations
Keywords: Urinary Incontinence, Stress; Tissue Therapy (Cell Therapy)
MeSH Terms: conditions — Urinary Incontinence; Urination Disorders; Urologic Diseases; Lower Urinary Tract Symptoms; Urological Manifestations; Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AMDC-USR (Experimental): Cell treatment
  Interventions: Biological: autologous muscle-derived cells (AMDC)

INTERVENTIONS:
Biological: autologous muscle-derived cells (AMDC) — Cell treatment

SUMMARY:
To study the safety and potential efficacy of Autologous Muscle Derived Cells for Urinary Sphincter Repair (AMDC-USR) for the treatment of male stress urinary incontinence (SUI) for patients that have undergone prior prostate surgery.

DETAILED DESCRIPTION:
This preliminary, prospective, single-arm clinical study will evaluate the safety and potential efficacy of Autologous Muscle Derived Cells for Urinary Sphincter Repair (AMDC-USR) for the treatment of male stress urinary incontinence (SUI) that develops following prostate surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male, at least 18 years old, with primary symptoms of SUI following prostate surgery,
* Patient has undergone prostate surgery but has not undergone radiation therapy, cryotherapy, or high-intensity focused ultrasound of the prostate,
* SUI severity should be ≥10 g and <400 g of urine leakage over 24 hours,
* Patient has failed to achieve acceptable resolution of SUI symptoms following prior therapy.

Exclusion Criteria:

* Symptoms of only urge urinary incontinence,
* Symptoms of stress urinary incontinence prior to prostate surgery,
* Routinely has more than 2 episodes of awakening to void during normal sleeping hours,
* Compromised immune system due to disease state, chronic corticosteroid use, or other immunosuppressive therapy,
* Previously treated with a periurethral balloon or adjustable sling for urinary incontinence,
* Symptoms of overflow incontinence
* Additional medical restrictions as specified in the Clinical Investigation Plan,
* Additional anatomical restrictions as specified in the Clinical Investigation Plan.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-02-19 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Peters, MD, Principal Investigator — Beaumont Hospital
Locations (5):
- United States (5):
  - University of Miami School of Medicine, Miami, Florida
  - Emory University Hospital, Atlanta, Georgia
  - William Beaumont Hospital, Royal Oak, Michigan
  - McKay Urology, Charlotte, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- AMDC-USR: Single intraurethral injection of 150 x 10^6 Autologous Muscle-Derived Cells (AMDCs)
Period: Overall Study
Arm/Group | AMDC-USR
Started | 25
Muscle Biopsy | 25
AMDC Injection | 23
1-Month Follow Up | 23
3-Month Follow Up | 23
6-Month Follow Up | 23
12-Month Follow Up | 23
Completed | 23
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | AMDC-USR
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 17
Age, Continuous [Median (Full Range); unit: years] | 67 [49 to 78]
Age, Customized [Mean (Standard Deviation); unit: years]
  Participant Age | 67.2 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25
Urinary Incontinence Type [Count of Participants; unit: Participants]
  Pure Stress Urinary Incontinence | 4
  Mixed Urinary Incontinence, Stress Predominant | 17
  Mixed Urinary Incontinence, Urge Predominant | 4
24-hour Pad Test Weight [Median (Full Range); unit: grams] — A test in which the participant wears specific absorbent pads dispensed by the clinic. The pads are weighed to record the pre-test weight prior to dispensing to the participant. The participant must wear the absorbent pads for 24 hours. The participant returns the used absorbent pads to the clinic, and the clinic records the post-test weight to determine urinary leakage for the 24 hour period. The difference in weights represent the amount of urine leaked.
  grams | 109.1 [4.1 to 431]
Incontinence Quality of Life (I-QOL) [Median (Full Range); unit: scores on scales] — The I-QOL questionnaire was a validated, 22-item tool used to assess QOL of participants with urinary incontinence. Scored 0 to 100, with higher scores indicating a better QOL.
  scores on scales | 59.1 [0 to 87.5]
International Consultation on Incontinence Questionnaire (ICIQ) [Median (Full Range); unit: scores on scales] — The ICIQ questionnaire was a validated 4-item tool used to assess symptom severity of participants with urinary incontinence. Scored 0 to 21, with lower scores indicating a better symptom severity.
  scores on scales | 13 [7 to 18]
International Prostate Symptom Score (IPSS) [Median (Full Range); unit: scores on scales] — The I-PSS was a validated questionnaire used to assess the severity of three urine storage symptoms (frequency, nocturia, urgency), four voiding symptoms (feeling of incomplete emptying, intermittency, straining, and a weak stream) and the degree of bother associated with those symptoms. A score of 0 to 7 indicates mild symptoms, 8 to 19 indicates moderate symptoms, and 20 to 35 indicates severe symptoms.
  scores on scales | 9 [1 to 33]
International Index of Erectile Function (IIEF) [Median (Full Range); unit: scores on scales] — The IIEF-5 questionnaire was a validated 5-item tool used to assess to presence and severity of erectile dysfunction (ED). Scored from 5 to 25, with lower scores indicating less ED symptoms.
  scores on scales | 13 [5 to 25]
Patient Global Impression of Severity (PGI-S) Questionnaire [Count of Participants; unit: Participants] — The PGI-S was a global assessment of symptom severity compared with severity before treatment started. Ratings that could be selected were: 1-normal, 2-mild, 3-moderate, and 4-severe.
  Participants
    Normal | 0
    Mild | 8
    Moderate | 13
    Severe | 4

OUTCOME MEASURES:

1. Primary Outcome: Rate of Product-related, Biopsy Procedure-related, and Injection Procedure-related Adverse Events
Description: Safety of AMDC-USR following treatment of SUI in male patients who have undergone prior prostate surgery was determined by the frequency and severity of adverse events related to study procedures and study product through 24 months following treatment of SUI in male patients who have undergone prior prostate surgery.
Time Frame: 24 months
Population: All subjects enrolled (biopsied)
Measure: Number; unit: events
Arm/Group | AMDC-USR
Number analyzed (Participants) | 25
events
  Study product-related serious adverse events | 0
  Study Product-related adverse events | 2
  Injection procedure-related adverse events | 0
  Biopsy procedure-related adverse events | 12

2. Primary Outcome: Volume of Post-void Residual (PVR) Urine
Description: Post void residual volume (PVR) was assessed through 12 months post-treatment to monitor potential retention or obstruction.
Time Frame: 1, 3, 6, and 12 months
Population: All subjects injected
Measure: Median (Full Range); unit: millileters
Arm/Group | AMDC-USR
Number analyzed (Participants) | 23
millileters
  Post void residual volume 1 month | 0 [0 to 52]
  Post void residual volume 3 months | 0 [0 to 37]
  Post void residual volume 6 months | 0 [0 to 142]
  Post void residual volume 12 months | 0 [0 to 22]

3. Secondary Outcome: Change From Baseline in Amount of Urine Leakage (Median 24 Hour Pad Weight)
Description: Change in the amount of urine leakage from baseline was assessed by 24-hour pad test at 1, 3, 6, and 12 months post-treatment. Amount of urine leakage experienced by subject at home during a 24-hour period; all pads used during test period are weighed before and after use and differences in weights represent the amount of urine leaked.
Time Frame: 1, 3, 6, and 12 months
Population: All subjects injected
Measure: Median (Full Range); unit: grams
Arm/Group | AMDC-USR
Number analyzed (Participants) | 23
grams
  24 hour pad weight at 1 month | 101.2 [5.3 to 674.3]
  24 hour pad weight at 3 months | 59.5 [18.1 to 357]
  24 hour pad weight at 6 months | 104.9 [9.2 to 359.5]
  24 hour pad weight at 12 months | 85.7 [13.5 to 319.7]

4. Secondary Outcome: Number of Participants With a Change From Baseline in Amount of Urine Leakage (Categorial ≥50% Reduction in 24-hour Pad Weight)
Description: Change in the amount of urine leakage from baseline was assessed by a 24-hour pad test at 1, 3, 6, and 12 months post-treatment. Amount of urine leakage experienced by subject at home during a 24-hour period; all pads used during test period are weighed before and after use and differences in weights represent the amount of urine leaked.
Time Frame: 1, 3, 6, and 12 months
Population: All subjects injected
Measure: Count of Participants; unit: Participants
Arm/Group | AMDC-USR
Number analyzed (Participants) | 23
Participants
  ≥50% reduction in 24 hour pad weight at 1 month | 2
  ≥50% reduction in 24 hour pad weight at 3 months | 4
  ≥50% reduction in 24 hour pad weight at 6 months | 4
  ≥50% reduction in 24 hour pad weight at 12 months | 7

5. Secondary Outcome: Median Change From Baseline in Patient-reported Quality of Life (QOL) - Incontinence Quality of Life (I-QOL) Questionnaire
Description: Median change from baseline in patient-reported quality of life (QOL) was assessed by the Incontinence Quality of Life (I-QOL) questionnaire at 1, 3, 6 and 12 months post-treatment. The I-QOL questionnaire was a validated, 22-item tool used to assess QOL of participants with urinary incontinence. Scored 0 to100, with higher scores indicating a better QOL.
Time Frame: 1, 3, 6, and 12 months
Population: All subjects injected
Measure: Median (Full Range); unit: points
Arm/Group | AMDC-USR
Number analyzed (Participants) | 23
points
  Change in I-QOL total score at 1 month | -6.8 [-14.8 to 6.8]
  Change in I-QOL total score at 3 months | 0 [-27.3 to 9.1]
  Change in I-QOL total score at 6 months | -9.1 [-37.5 to 12.5]
  Change in I-QOL total score at 12 months | -9.1 [-36.4 to 14.8]

6. Secondary Outcome: Median Change From Baseline in Patient-reported Symptom Severity- International Consultation on Incontinence Questionnaire (ICIQ)
Description: Median change from baseline in patient-reported symptom severity was assessed by the International Consultation on Incontinence Questionnaire (ICIQ) questionnaire at 1, 3, 6, and 12 months post-treatment. The ICIQ questionnaire was a validated 4-item tool used to assess symptom severity of participants with urinary incontinence. Scored 0 to 21, with lower scores indicating a better symptom severity.
Time Frame: Baseline, 1, 3, 6, and 12 months
Population: All subjects injected
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | AMDC-USR
Number analyzed (Participants) | 23
scores on a scale
  Change in ICIQ score at 1 month | 0 [-2 to 7]
  Change in ICIQ score at 3 months | 0 [-3 to 7]
  Change in ICIQ score at 6 months | 0 [-3 to 7]
  Change in ICIQ score at 12 months | 1 [-1 to 16]

7. Secondary Outcome: Median Change in Patient-reported Incontinence Symptom Severity - International Prostate Symptom Score (I-PSS) Questionnaire
Description: Patient-reported incontinence symptom severity was assessed by questionnaires at 1, 3, 6, and 12 months post-treatment using the International Prostate Symptom Score (I-PSS) questionnaire. The I-PSS was a validated questionnaire used to assess the severity of three urine storage symptoms (frequency, nocturia, urgency), four voiding symptoms (feeling of incomplete emptying, intermittency, straining, and a weak stream) and the degree of bother associated with those symptoms. A score of 0 to 7 indicates mild symptoms, 8 to 19 indicates moderate symptoms, and 20 to 35 indicates severe symptoms.
Time Frame: Baseline, 1, 3, 6, and 12 months
Population: All subjects injected
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | AMDC-USR
Number analyzed (Participants) | 23
scores on a scale
  Change in I-PSS score at 1 month | 1 [-4 to 8]
  Change in I-PSS score at 3 months | 1 [-8 to 10]
  Change in I-PSS score at 6 months | 1 [-6 to 15]
  Change in I-PSS score at 12 months | 1 [-3 to 10]

8. Secondary Outcome: Distribution of Patient-reported Incontinence Symptom Severity Scores - Patient Global Impression of Severity (PGI-S) Questionnaire
Description: Patient-reported incontinence symptom severity was assessed by questionnaires at 1, 3, 6, and 12 months post-treatment using the Patient Global Impression of Severity (PGI-S) questionnaire. The PGI-S was a global assessment of symptom severity compared with severity before treatment started. Ratings that could be selected were: 1-normal, 2-mild, 3-moderate, and 4-severe. Percentages of participants in each category were determined at each visit.
Time Frame: 1, 3, 6, and 12 months
Population: All subjects injected
Measure: Count of Participants; unit: Participants
Arm/Group | AMDC-USR
Number analyzed (Participants) | 23
Participants
  PGI-S score at 1 month: Normal | 1
  PGI-S score at 1 month: Mild | 3
  PGI-S score at 1 month: Moderate | 13
  PGI-S score at 1 month: Severe | 6
  PGI-S score at 3 months: Normal | 0
  PGI-S score at 3 months: Mild | 8
  PGI-S score at 3 months: Moderate | 12
  PGI-S score at 3 months: Severe | 3
  PGI-S score at 6 months: Normal | 0
  PGI-S score at 6 months: Mild | 9
  PGI-S score at 6 months: Moderate | 11
  PGI-S score at 6 months: Severe | 3
  PGI-S score at 12 months: Normal | 1
  PGI-S score at 12 months: Mild | 6
  PGI-S score at 12 months: Moderate | 13
  PGI-S score at 12 months: Severe | 3

9. Secondary Outcome: Distribution of Patient-reported Incontinence Symptom Severity Scores - Patient Global Impression of Improvement (PGI-I) Questionnaire
Description: Patient-reported incontinence symptom severity was assessed by questionnaires at 1, 3, 6, and 12 months post-treatment using the Patient Global Impression of Improvement (PGI-I) questionnaire. The PGI-I was a global assessment of symptom severity in which participants selected the following ratings: 1-Very much better, 2-Much better, 3-A little better, 4-No change, 5-A little worse, 6-Much worse, and 7-Very much worse. Percentages of participants in each category were determined at each visit.
Time Frame: 1, 3, 6, and 12 months
Population: All subjects injected
Measure: Count of Participants; unit: Participants
Arm/Group | AMDC-USR
Number analyzed (Participants) | 23
Participants
  PGI-I score at 1 month: Very much better | 1
  PGI-I score at 1 month: Much better | 0
  PGI-I score at 1 month: A little better | 4
  PGI-I score at 1 month: No change | 18
  PGI-I score at 1 month: A little worse | 0
  PGI-I score at 3 months: Very much better | 0
  PGI-I score at 3 months: Much better | 1
  PGI-I score at 3 months: A little better | 12
  PGI-I score at 3 months: No change | 9
  PGI-I score at 3 months: A little worse | 1
  PGI-I score at 6 months: Very much better | 0
  PGI-I score at 6 months: Much better | 3
  PGI-I score at 6 months: A little better | 11
  PGI-I score at 6 months: No change | 7
  PGI-I score at 6 months: A little worse | 2
  PGI-I score at 12 months: Very much better | 0
  PGI-I score at 12 months: Much better | 4
  PGI-I score at 12 months: A little better | 11
  PGI-I score at 12 months: No change | 5
  PGI-I score at 12 months: A little worse | 3

10. Secondary Outcome: Median Change From Baseline in Patient-reported Erectile Dysfunction (ED) - Index of Erectile Function (IIEF-5) Questionnaire
Description: SUI and ED can be comorbidities that develop following prostate surgery; median change from baseline in patient-reported Erectile Dysfunction (ED) was assessed by the 5-Item International Index of Erectile Function (IIEF-5). The IIEF-5 questionnaire was a validated 5-item tool used to assess to presence and severity of erectile dysfunction. Scored from 5 to 25, with lower scores indicating less ED symptoms.
Time Frame: Baseline, 1, 3, 6, and 12 months
Population: All subjects injected
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | AMDC-USR
Number analyzed (Participants) | 23
scores on a scale
  Change in IEEF-5 score at 1 month | 0 [-9 to 8]
  Change in IEEF-5 score at 3 months | 0 [-7 to 8]
  Change in IEEF-5 score at 6 months | 0 [-11 to 4]
  Change in IEEF-5 score at 12 months | 0 [-8 to 7]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from enrollment through study exit - 24 months total.
Description: All adverse events were collected at baseline, 1 month, 3 months, 6 months, 12 months, and 24 months post-treatment. Any adverse events occurring in ≥ 5% of participants are reported. Adverse events assessed as AMDC product-related or biopsy procedure-related were reported regardless of frequency threshold. No injection procedure-related adverse events were reported.
Arm/Group | AMDC-USR
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 4/25
Other Adverse Events (participants affected / at risk) | 9/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AMDC-USR (N=25)
Myocardial infarction (Cardiac disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AMDC-USR (N=25)
Micturition urgency (Renal and urinary disorders) | 1 (1) — Study Product-Related Adverse Event
Pollakiuria (Renal and urinary disorders) | 1 (1) — Study Product-Related Adverse Event
Post procedural contusion (Injury, poisoning and procedural complications) | 2 (2) — Biopsy Procedure-Related Adverse Event, AEs with ≥5% Frequency
Post procedural swelling (Injury, poisoning and procedural complications) | 1 (1) — Biopsy Procedure-Related Adverse Event
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (1) — Biopsy Procedure-Related Adverse Event
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1) — Biopsy Procedure-Related Adverse Event
Procedural pain (Injury, poisoning and procedural complications) | 3 (3) — Biopsy Procedure-Related Adverse Event, AEs with ≥5% Frequency
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) — 1 Event Biopsy Procedure-Related Adverse Event, 1 Event Not Related to Study Product or Procedures, AEs with ≥5% Frequency
Hypoaesthesia (Nervous system disorders) | 1 (1) — Biopsy Procedure-Related Adverse Event
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) — Biopsy Procedure-Related Adverse Event
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) — Biopsy Procedure-Related Adverse Event
Abdominal Pain (Gastrointestinal disorders) | 2 (2) — AEs Not Related to Study Product or Procedures with ≥5% Frequency
Sinusitis (Infections and infestations) | 2 (7) — AEs Not Related to Study Product or Procedures with ≥5% Frequency
Fall (Injury, poisoning and procedural complications) | 2 (2) — AEs Not Related to Study Product or Procedures with ≥5% Frequency
Laceration (Infections and infestations) | 2 (2) — AEs Not Related to Study Product or Procedures with ≥5% Frequency

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-17): https://cdn.clinicaltrials.gov/large-docs/32/NCT02291432/Prot_SAP_000.pdf